CLINICAL TRIAL: NCT05066438
Title: The Effect of Prenatal Hand Expression on the Rate of Exclusive Breastfeeding to Two Months
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Almereau Prollius, Principal Investigator, University of Saskatchewan
Other Study IDs: Bio 2238
Record Dates: First submitted 2021-09-21; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Breastfeeding; Breastfeeding, Exclusive; Breast Milk Collection
Keywords: antenatal; colostrum; hand expression; prenatal
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antenatal hand expression - intention to exclusively breastfeed: Eligible participants in this group intend to exclusively breastfeed AND must have received standardized counselling on and practiced antenatal hand expression for a minimum of 10 days beginning no earlier than 36 weeks gestational age.
  Interventions: Behavioral: Antenatal hand expression
- No antenatal hand expression - intention to exclusively breastfeed: Eligible participants in this group intend to exclusively breastfeed but have NOT received any standardized counselling on antenatal hand expression and have not practiced antenatal hand expression OR have practiced antenatal hand expression but for less than 10 days.

INTERVENTIONS:
Behavioral: Antenatal hand expression — Standardized counselling and provision of information/resources on the practice of antenatal hand expression to encourage milk let down and colostrum production/collection.
  Groups: Antenatal hand expression - intention to exclusively breastfeed

SUMMARY:
Despite recommendations by several health authorities, the rate of sustained exclusive breastfeeding for two months is less than fifty-five percent in Canada. The two most common reasons for early discontinuation are problems with milk supply and difficulty with technique. Antenatal hand expression (AHE) is a method used to assist with colostrum collection in low-risk pregnancies near term. This method has been shown to have several benefits, including increased milk supply at birth. This study aims to determine if the employment of antenatal hand expression in low-risk pregnancies near term affects the rate of sustained breastfeeding exclusively to two months.

ELIGIBILITY:
Inclusion Criteria:

* inclusion to breastfeed
* no contraindications to vaginal delivery
* multiple gestation only if cleared for vaginal delivery

Exclusion Criteria:

* intention to formula feed
* antenatal hand expression training provided by staff outside of study protocol
* practiced antenatal hand expression prior to 36 weeks gestation
* breech presentation
* history of preterm labour, preterm birth or threatened preterm labour
* history of (or current) cervical insufficiency
* any contraindication to vaginal delivery (ie. placenta or vasa previa, classical uterine scar, etc.)
* intrauterine growth restriction
* antepartum hemorrhage
* any contraindication to breastfeeding (eg. HIV)
* multiple gestation requiring Cesarean delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women in Saskatoon, Saskatchewan who intend to breastfeed. Prospective participants will be invited to enrol in this study if they meet inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Exclusive breastfeeding to two months | This metric measured by questionnaire at two months
  Participant-reported data on newborn dietary intake, collected by telephone questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Almereau Prollius, MD, Principal Investigator — University of Saskatchewan

IPD SHARING:
Plan to Share IPD: No